CLINICAL TRIAL: NCT03235921
Title: Use of Nitroglycerine to Improve Signs of Poor Peripheral Perfusion in Patients With Traumatic Hemorrhagic Shock
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, medhat sayed ali, Resident at Anaesthesia, ICU and pain management department,Assiut University, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15316
Record Dates: First submitted 2016-08-19; First posted 2017-08-01 (Actual); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Hemorrhagic Shock
Keywords: hemorrhagic shock; perfusion index; lactate; nitroglycerin
MeSH Terms: conditions — Shock, Hemorrhagic | interventions — Nitroglycerin

STUDY DESIGN:
Intervention Model Description: To avoid significant hypotension during nitroglycerin administration, each patient was evaluated for adequate intravascularvolume as evidenced by repeated volume challenges(250 mL of crystalloid over 10 minutes) up to appoint at which central venous pressure raised by more than 2 mmHg.
  When the systolic blood pressure reaches 90mmHg or more we can apply the nitroglycerin patch of 2.5 mg alongside with continuous resuscitation the dose can be doubled according to the change in the peripheral perfusion parameters. Time between administration of nitroglycerin patch and peak of its action will be calculated.
  Nitroglycerin patch will be removed if the patient developed significant hypotension (mean arterial pressure of less than 50 mm Hg ) however its action may persist up to 45minutes after removal.
  During the study, infusion rates of noradrenaline or other vasoactive drugs were not changed and no additional fluids were administered.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- nitroglycerin (Other): nitroglycerin patch 5 mg applied to front of chest in each patient at time of admission once.
  Interventions: Drug: Nitroglycerin patch 5mg
- control group (Other): no drug given to the patients in control group
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Nitroglycerin patch 5mg — application of the nitroglycerin patch 5 mg to each patient in nitroglycerin group
  Other Names: nitroglycerin
  Arms: nitroglycerin
Other: placebo — no drug given to the control group
  Arms: control group

SUMMARY:
Hemorrhagic shock is a pathologic state in which intravascular volume and oxygen delivery are impaired. During circulatory failure associated with hypovolemia and low cardiac output, redistribution of blood flow caused by increased vasoconstriction results in decreased perfusion of the skin.

Skin temperature and capillary refill time has been advocated as a measure of peripheral perfusion.

DETAILED DESCRIPTION:
Perfusion index (PI) is a non-invasive numerical value of peripheral perfusion obtained from pulse oximetry, it is an indicator of the pulse strength at the sensor site. The PI's values range from 0.2% for very weak pulse to 20% for extremely strong pulse according to patient's physiological conditions and monitoring sites.

Large increases in lactate (i.e. > 5 mmol/L) usually only occur due to hypoperfusion or muscle activity such as exercise or seizures.

This study will investigate the role of nitroglycerine patch in improving the peripheral perfusion in poly traumatized patient with hemorrhagic shock for the first time.

ELIGIBILITY:
Inclusion Criteria:

* Age: 20-60 years old. With the patient fully conscious or slightly drowsy.
* Blood pressure: Systolic blood pressure below 90mmhg ,mean blood pressure below70mmhg or decrease of systolic blood pressure 40mmhg below normal value.
* Metabolic acidosis: PH less than 7.35 due to hypoperfusion.
* Capillary refill time > 4 seconds.
* Normal body core temperature.

Exclusion Criteria:

* Age: below 20 and above 60 years old.
* Head trauma with Glasco coma score below 14 due to increased intracranial pressure (stroke, subarachnoid hemorrhage or brain trauma injury).
* Severe hypotension not responding to fluid therapy.
* Patient with bilateral ischemic arm injury.
* Patient with hepatic cell failure
* Patients admitted to the emergency trauma department after 6 hours of the trauma event.
* Preexisting conditions as severe cardiovascular disease, uncontrolled hemorrhage, failure of central venous catheterization, dialytic procedure anticipated during the study period.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-08 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
increase of perfusion index PI measured by pulse oximeter | 48hours
  nitroglycerin increases the perfusion index in patients with hemorrhagic shock more than in control group without use of nitroglycerin

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Kotb, professor, Principal Investigator — assuit university faculty of medicine
Locations (1):
- Assuit University Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Kauvar DS, Wade CE. The epidemiology and modern management of traumatic hemorrhage: US and international perspectives. Crit Care. 2005;9 Suppl 5(Suppl 5):S1-9. doi: 10.1186/cc3779. Epub 2005 Oct 7. PMID 16221313
- [Background] Bond RF. A review of the skin and muscle hemodynamics during hemorrhagic hypotension and shock. Adv Shock Res. 1982;8:53-70. PMID 6753542
- [Background] Schriger DL, Baraff LJ. Capillary refill--is it a useful predictor of hypovolemic states? Ann Emerg Med. 1991 Jun;20(6):601-5. doi: 10.1016/s0196-0644(05)82375-3. PMID 2039096
- [Background] Steiner MJ, DeWalt DA, Byerley JS. Is this child dehydrated? JAMA. 2004 Jun 9;291(22):2746-54. doi: 10.1001/jama.291.22.2746. PMID 15187057
- [Background] Vincent JL, Ince C, Bakker J. Clinical review: Circulatory shock--an update: a tribute to Professor Max Harry Weil. Crit Care. 2012 Nov 20;16(6):239. doi: 10.1186/cc11510. PMID 23171699
- [Background] Lima AP, Beelen P, Bakker J. Use of a peripheral perfusion index derived from the pulse oximetry signal as a noninvasive indicator of perfusion. Crit Care Med. 2002 Jun;30(6):1210-3. doi: 10.1097/00003246-200206000-00006. PMID 12072670
- [Background] Gladden LB. Lactate metabolism: a new paradigm for the third millennium. J Physiol. 2004 Jul 1;558(Pt 1):5-30. doi: 10.1113/jphysiol.2003.058701. Epub 2004 May 6. PMID 15131240
- [Background] Lopez A, Lorente JA, Steingrub J, Bakker J, McLuckie A, Willatts S, Brockway M, Anzueto A, Holzapfel L, Breen D, Silverman MS, Takala J, Donaldson J, Arneson C, Grove G, Grossman S, Grover R. Multiple-center, randomized, placebo-controlled, double-blind study of the nitric oxide synthase inhibitor 546C88: effect on survival in patients with septic shock. Crit Care Med. 2004 Jan;32(1):21-30. doi: 10.1097/01.CCM.0000105581.01815.C6. PMID 14707556
- [Background] Vincent JL, Zhang H, Szabo C, Preiser JC. Effects of nitric oxide in septic shock. Am J Respir Crit Care Med. 2000 Jun;161(6):1781-5. doi: 10.1164/ajrccm.161.6.9812004. PMID 10852744
- [Background] LILLEHEI RC, LONGERBEAM JK, BLOCH JH, MANAX WG. THE NATURE OF IRREVERSIBLE SHOCK: EXPERIMENTAL AND CLINICAL OBSERVATIONS. Ann Surg. 1964 Oct;160(4):682-710. doi: 10.1097/00000658-196410000-00012. No abstract available. PMID 14210369
- [Background] Nguyen HB, Loomba M, Yang JJ, Jacobsen G, Shah K, Otero RM, Suarez A, Parekh H, Jaehne A, Rivers EP. Early lactate clearance is associated with biomarkers of inflammation, coagulation, apoptosis, organ dysfunction and mortality in severe sepsis and septic shock. J Inflamm (Lond). 2010 Jan 28;7:6. doi: 10.1186/1476-9255-7-6. PMID 20181046
- [Background] SpO2 Monitors with OXISMART® Advanced Signal Processing and Alarm Management Technology. Pulse Oximetry Note Number 9. Masimo signal extraction technology 2008.
- [Background] American College of Surgeons Committee on Trauma: Advanced TraumaLife Support for Doctors: Instructor Course Manual. 8th ed. Chicago, Ill: AmericanCollege of Surgeons; 2008.